CLINICAL TRIAL: NCT03090321
Title: MyHeart Counts Cardiovascular Health Study
Acronym: MHC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Euan Ashley, Associate Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 31409
Record Dates: First submitted 2016-12-14; First posted 2017-03-24 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-03

CONDITIONS: Cardiovascular Health
Keywords: fitness; health; activity; heart risk; wellness
MeSH Terms: conditions — Motor Activity | interventions — acetohydroxamic acid

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (5):
- Stand Prompt (Active Comparator): Behavioral Intervention Prompt- Participant will receive a notification asking them to stand and walk if they have been sitting for longer than 60 minutes.
  Interventions: Behavioral: Stand Prompt
- Step Prompt (Active Comparator): The participant will receive a notification if they are below 5000 steps by 3pm each day asking them to get to 10000 steps.
  Interventions: Behavioral: Step Prompt
- Cluster Prompt (Active Comparator): The participant will receive daily information notifications specific to the activity cluster they fall into based on the activity data collected in phase 1 of the study.
  Interventions: Behavioral: Cluster Prompt
- Read AHA website (Placebo Comparator): Daily reminder to read the American Heart Association (AHA) website.
  Interventions: Behavioral: Read AHA website
- Baseline monitoring (No Intervention): No feedback is provided to the users. This is the control arm.

INTERVENTIONS:
Behavioral: Stand Prompt — The participant will receive a notification asking them to stand or walk if they have been sitting for longer than 60 minutes
  Other Names: Behavior Change and Motivational Coaching-Stand Prompt
  Arms: Stand Prompt
Behavioral: Step Prompt — The participant will receive a notification if they are below 5000 steps by 3pm each day asking them to get to 10000 steps.
  Other Names: Behavior Change and Motivational Coaching- Step Prompt
  Arms: Step Prompt
Behavioral: Cluster Prompt — The participant will receive daily information notifications specific to the activity cluster they fall into based on the activity data collected in phase 1 of the study
  Other Names: Behavior Change and Motivational Coaching- Cluster Prompt
  Arms: Cluster Prompt
Behavioral: Read AHA website — Daily reminder to read the newsfeed from the American Heart Association (AHA) website, this is a control arm
  Other Names: Behaviour Change and Motivational Coaching- Reminder to read the American Heart Association (AHA) website
  Arms: Read AHA website

SUMMARY:
The MyHeart Counts Cardiovascular Health Study will utilize mobile health capabilities of smartphones and wearables to assess daily activity measures of the general population and compare these to measures of cardiovascular health risk factors and fitness. How people divide their time among exercise, sedentary behavior, and sleep all affect cardiovascular health, yet to date these have largely gone unmeasured. With the advancement of phone sensors and wearable fitness tracking devices these factors are now more straightforward to gather and measure. The use of smartphones by a large segment of the population allows for data collection on an unprecedented scale. The investigators aim to amass activity and cardiovascular health data on thousands of participants as well as provide significantly more quantitative data on type,duration, and intensity of daily activities.

In the second phase of the MyHeart Counts Cardiovascular Health Study (Randomized Assessment of Physical Activity Prompts In A Large Ambulatory Population) the researchers will conduct a randomized controlled clinical trial of four different physical activity prompts (intervention) and their effect on the level of physical activity in the study population as measured by change in step count.

DETAILED DESCRIPTION:
MyHeart Counts Cardiovascular Health Study is a smartphone-based mobile cardiovascular health research study. The study will utilize the mobile health capabilities of smartphones and wearables to assess daily activity measures of the general public and compare these to measures of cardiovascular health - risk factors and fitness. How people divide their time among exercise, sedentary behavior, and sleep all affect cardiovascular health, yet these largely go unmeasured. With the advancement in phone sensors and wearables these factors are now more straightforward to gather and measure. The use of smartphones by a large segment of the population allows for data collection on an unprecedented scale. The investigators aim to amass activity and cardiovascular health data on thousands of participants as well as provide much more quantitative data on type,duration, and intensity of daily activities. The MyHeart Counts Cardiovascular Health mobile application provides a platform for the investigation of methods aimed to aid participants in increasing heart healthy activities. The overall goal of the study is to develop an extensive source of data which will inform future cardiovascular health guidelines.

In the second phase of the MyHeart Counts Cardiovascular Health Study (Randomized Assessment of Physical Activity Prompts In A Large Ambulatory Population) the investigators will conduct a randomized controlled clinical trial of four different physical activity prompts (intervention) and their effect on increasing physical activity in the study population as measured by change in step count.

Of note to supplement the activity data the investigators will ask participants who have completed a genetic analysis to share their that data with the MyHeart Counts Cardiovascular Health Study research team. The investigators believe the opportunity to overlay activity, heart risk and genetic data for participants is a great tool for discovery.

ELIGIBILITY:
Inclusion Criteria:

* All adults over the age of 18

Exclusion Criteria:

* Children under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000000 (Estimated)
Dates: Start 2015-03; Primary Completion 2026-07 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Activity frequency and duration as Measured By Smartphone Core Motion Chip Sensor (Step count as seen in Apple's Healthkit) | 5 weeks
  The researchers will compare step count data collected during baseline (or phase 1) week with step count data at the end of each of the 4 intervention weeks.

SECONDARY OUTCOMES:
Change in self reported levels of happiness as indicated on a numerical gradient scale and self reported by participant using the OECD Guidelines on Measuring Subjective Well Being survey | 5 weeks
Change in responses ( to survey questions on self perceived risk of cardiovascular disease and well being (survey adopted from reference in description) | 5 weeks
  Each answer prompt on the survey is given a unique numerical value which is then added and averaged. The researchers will investigate for changes in this score at baseline and during interventions.
Change in sleep duration as measured by Apples core motion chip. | 5 weeks
  The iphone is able to track sleep by sensing lack of motion between self reported sleeping and wake times. The investigators will compare the average sleep time detected by phone at baseline and at the end of each intervention week.
Change in self reported sleep duration obtained from a daily user survey. | 5 weeks
  The researchers will compare self reported sleep time at baseline vs end of each intervention week.

CONTACTS AND LOCATIONS:
Overall Officials: Euan Ashley, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual user data will not be shared, deidentified user data will be shared if the user has indicated that this is ok with them.

REFERENCES:
- [Background] Organisation for Economic Co-operation and Development (OECD). OECD Guidelines on Measuring Subjective Well-being. Paris: OECD Publishing; 2013 Mar 20. Available from http://www.ncbi.nlm.nih.gov/books/NBK189560/ PMID 24600748
- [Background] Knowles JW, Assimes TL, Kiernan M, Pavlovic A, Goldstein BA, Yank V, McConnell MV, Absher D, Bustamante C, Ashley EA, Ioannidis JP. Randomized trial of personal genomics for preventive cardiology: design and challenges. Circ Cardiovasc Genet. 2012 Jun;5(3):368-76. doi: 10.1161/CIRCGENETICS.112.962746. No abstract available. PMID 22715281
- [Background] Hershman SG, Bot BM, Shcherbina A, Doerr M, Moayedi Y, Pavlovic A, Waggott D, Cho MK, Rosenberger ME, Haskell WL, Myers J, Champagne MA, Mignot E, Salvi D, Landray M, Tarassenko L, Harrington RA, Yeung AC, McConnell MV, Ashley EA. Physical activity, sleep and cardiovascular health data for 50,000 individuals from the MyHeart Counts Study. Sci Data. 2019 Apr 11;6(1):24. doi: 10.1038/s41597-019-0016-7. PMID 30975992
- [Background] McConnell MV, Shcherbina A, Pavlovic A, Homburger JR, Goldfeder RL, Waggot D, Cho MK, Rosenberger ME, Haskell WL, Myers J, Champagne MA, Mignot E, Landray M, Tarassenko L, Harrington RA, Yeung AC, Ashley EA. Feasibility of Obtaining Measures of Lifestyle From a Smartphone App: The MyHeart Counts Cardiovascular Health Study. JAMA Cardiol. 2017 Jan 1;2(1):67-76. doi: 10.1001/jamacardio.2016.4395. PMID 27973671
- [Background] Shcherbina A, Hershman SG, Lazzeroni L, King AC, O'Sullivan JW, Hekler E, Moayedi Y, Pavlovic A, Waggott D, Sharma A, Yeung A, Christle JW, Wheeler MT, McConnell MV, Harrington RA, Ashley EA. The effect of digital physical activity interventions on daily step count: a randomised controlled crossover substudy of the MyHeart Counts Cardiovascular Health Study. Lancet Digit Health. 2019 Nov;1(7):e344-e352. doi: 10.1016/S2589-7500(19)30129-3. Epub 2019 Oct 9. PMID 33323209
- [Derived] Javed A, Kim DS, Hershman SG, Shcherbina A, Johnson A, Tolas A, O'Sullivan JW, McConnell MV, Lazzeroni L, King AC, Christle JW, Oppezzo M, Mattsson CM, Harrington RA, Wheeler MT, Ashley EA. Personalized digital behaviour interventions increase short-term physical activity: a randomized control crossover trial substudy of the MyHeart Counts Cardiovascular Health Study. Eur Heart J Digit Health. 2023 Aug 9;4(5):411-419. doi: 10.1093/ehjdh/ztad047. eCollection 2023 Oct. PMID 37794870